CLINICAL TRIAL: NCT02868905
Title: Identification of Epigenetic Markers Common to Obesity and Alzheimer's Disease in Women - Pilot Study
Brief Title: Identification of Epigenetic Markers Common to Obesity and Alzheimer's Disease in Women
Acronym: Oba
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-A01686-43
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Obesity; Alzheimer's Disease
MeSH Terms: conditions — Obesity; Alzheimer Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control group (Other): Control group
  Interventions: Procedure: Blood sample
- Obese group (Other): Obese group
  Interventions: Procedure: Blood sample
- Non-obese AD group (Other): Non-obese AD groups
  Interventions: Procedure: Blood sample
- Obese AD group (Other): Obese AD group
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample

SUMMARY:
The purpose of this study is to compare average methylation of epigenetic markers on genomic DNA and some genes (APP, BACE, LRP, SorL1) involved in cerebral amyloid homeostasis:

* Of obese young adults and healthy young adults
* Of obese young adults and individuals affected by Alzheimer's disease (AD) having been obese at young adult age (<50 years old) or individuals affected by Alzheimer's disease (AD) having never been obese.

The secondary purpose is to determine if there is an association between the frequency of these epigenetic markers and elements associated to the metabolic syndrome (lipidic and glycemic analysis, leptinemia, inflammation markers) and clinical ones (visceral fat mass, body mass index) in young adults.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* 18-50 year old women, age- (10 years) and sociocultural-matched with group 2
* Non obese and never been obese
* 18.5 < BMI < 25
* Folstein MMS > 27
* Informed consent
* Affiliation to social security plan

Group 2:

* 18-50 year old women, age- (10 years) and sociocultural-matched with group 1
* Waist size > 88cm
* 30 < BMI < 45
* Insulin-resistant patients (Insulin resistance index, HOMA-IR > 3.8)
* Obesity onset during childhood (pre-puberty period)
* Folstein MMS > 27
* Informed consent
* Affiliation to social security plan

Group 3:

* >60 year old women, age- (10 years) matched with group 4
* No obesity history (18.5 ≤ BMI < 25 at adult age)
* Sporadic forms of mild to moderate AD with demonstration of AD physiopathologic process according to new recommendations of 2011 of National Institute on Aging and Alzheimer's Association on diagnostic guidelines for Alzheimer's disease
* 15< Folstein MMS ≤ 26
* Informed consent
* Affiliation to social security plan

Group 4:

* >60 year old women, age- (10 years) matched with group 3
* Obesity history (BMI > 30 at least one time at adult age)
* Sporadic forms of mild to moderate AD with demonstration of AD physiopathologic process according to new recommendations of 2011 of National Institute on Aging and Alzheimer's Association on diagnostic guidelines for Alzheimer's disease
* 15 < Folstein MMS ≤ 26
* Informed consent
* Affiliation to social security plan

Exclusion Criteria:

Group 1:

* <18
* Patient under guardianship, curatorship or judicial protection
* Folate supplementation
* Diabetic or glucose intolerant subjects
* Present participation to another study with neuropsychological evaluation and/or drug administration
* Pregnant women

Groups 2,3 and 4:

* <18
* Patient under guardianship, curatorship or judicial protection
* Folate supplementation
* Present participation to another study with neuropsychological evaluation and/or drug administration

Group 2:

- Pregnant women

Group 4:

- Obese or overweight patients (BMI>25)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Methylation of CpG islands in genomic DNA and in 4 target genes involved in AD (APP, SorLA/LR11, BACE1, LRP) in obese and AD subjects | day 0

SECONDARY OUTCOMES:
body mass index | day 0
visceral fat mass level | day 0
leptinemia by ELISA | day 0
insulinemia by ELISA | day 0
glycemia | day 0
triglyceridemia | day 0
HDL cholesterol level in blood | day 0
Reactive C protein level in blood | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Thérèse RIVASSEAU-JONVEAUX, Principal Investigator — Service de Gériatrie, Hôpitaux de Brabois, 3 rue du Morvan, 54 511 Vandoeuvre-lès-Nancy
Locations (1):
- CHRU de Nancy, Nancy, France